CLINICAL TRIAL: NCT05908864
Title: Efficacy of Nebulized Versus Intravenous Magnesium Sulfate in Treatment of Asthma Exacerbation
Brief Title: Nebulized Versus Intravenous Magnesium Sulfate in Treatment of Asthma Exacerbation
Status: Completed | Type: Observational
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Raghda R.S. Hussein, Assistant Professor of Clinical Pharmacy, Beni-Suef University
Other Study IDs: #FWA00015574
Record Dates: First submitted 2023-05-26; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Asthma Attack
MeSH Terms: interventions — Magnesium Sulfate

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- IV Magnesium Sulfate
  Interventions: Drug: Magnesium sulfate
- Inhaled Magnesium Sulfate
  Interventions: Drug: Magnesium sulfate
- Control group
  Interventions: Drug: Magnesium sulfate

INTERVENTIONS:
Drug: Magnesium sulfate — Blood pressure, respiratory rate, pulse, peak expiratory flow rate (PEFR) measurement using a peak flowmeter, Fischl index and need for hospitalization in patients with acute bronchial asthma were done

SUMMARY:
A prospective study in Beni-Seuf University Hospital that was conducted on 123 adult patients with acute asthma exacerbations. Patients were classified into group (I): received IV magnesium sulfate, group (II): received nebulized magnesium sulfate, and group (III): control group. Blood pressure, respiratory rate, pulse, peak expiratory flow rate (PEFR) measurement using a peak flowmeter, Fischl index and need for hospitalization in patients with acute bronchial asthma were done for all patients before treatment, immediately after the treatment, "30", and "60" min after treatment.

DETAILED DESCRIPTION:
Inclusion criteria :

* adult patients between the ages of 18 and 50 years with acute attack of bronchial asthma
* from both sexes
* Normal renal function
* Normal cardiovascular function

Exclusion criteria:

* Patients were younger than 18 years or older than 50 years.
* Patients suffered from chronic obstructive pulmonary disease, renal disorder and heart failure

All patients were subjected to: complete history taking, blood sampling for serum magnesium measurement (on admission before the initial treatment and after the initial treatment) the patients were randomly separated into 3 equal groups each group consists of 41 patients.

The 1ST group has been managed by an initial treatment plan (consists of supplemental oxygen therapy to keep oxygen saturation higher than 90%., nebulization of 1 ml salbutamol respirator solution mixed with 9 ml normal saline solution for one session [Farcolin respirator solution: each 20 ml of Farcolin contains Salbutamol sulfate 0.121 gm. Made in Egypt, by: Pharco Pharmaceuticals -Alexandria], Intravenous administration of hydrocortisone 100 mg for a single dose [Solu-Cortef: vial contains powder of 100 mg Sodium hydrocortisone sodium succinate dissolved with 2 ml solvent of sterile bacteriostatic water for IV injection. Manufactured by: Egyptian Int. Pharmaceutical Industries co. (e.i.p.i.co.) - Egypt. Under license of: Pfizer]) plus a single dose (2000 mg) of magnesium sulfate prepared by mixing 20 ml of 10 % magnesium sulfate (2000 MG) [14] ,manufactured by Memphis Pharmaceuticals and Chemical Industries, with 30 ml of distillated water for injection to produce 50 ml of isotonic magnesium sulfate solution (324 MSOM/L) administered intravenously over 1 hour.

The 2nd group has been managed by the same initial treatment plan plus a single dose (2000 mg) of magnesium sulfate prepared by mixing 20 ml of 10 % magnesium sulfate (2000 MG) [14] ,manufactured by Memphis Pharmaceuticals and Chemical Industries, with 30 ml of distillated water to produce 50 ml of isotonic magnesium sulfate solution (324 MSOM/L). nebulized using jet nebulizer over 1 hour.

The 3rd group has been managed by the same treatment plan Without using magnesium sulfate. (a control group) the following were recorded for each patient at a fixed interval (before the initial treatment, immediately after the initial treatment, 30, and 60 min after the initial treatment):

1. blood pressure, respiratory rate and pulse rate
2. Peak expiratory flow measurement using peak flow meter.
3. Fischl index for relapse and need for hospitalization in patients with acute bronchial asthma. [16[ .

ELIGIBILITY:
Inclusion Criteria:

* adult patients between the ages of 18 and 50 years with acute attack of bronchial asthma
* From both sexes
* Normal Renal function
* Normal Cardiovascular function

Exclusion Criteria:

* Patients were younger than 18 years or older than 50 years.
* Patients suffered from chronic obstructive pulmonary disease
* Patidnts suffered from renal disorder
* Patients with heart failure.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 131 patients were included in the study.Eight subjects were excluded due to presence of heart failure or renal failure.
Sampling Method: Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2019-11-22 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Improving pulmonary function tests as PEFR for asthmatic patients | 13 monthes
  Prevention of the progression asthma exacerbation for included subjects

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Beni-suef university, Banī Suwayf, Egypt

IPD SHARING:
Plan to Share IPD: No